CLINICAL TRIAL: NCT00652418
Title: Evaluation of a Single Intravenous Injection of Magnevist (SH L 451 A) at 0.1 mmol/kg and 0.2 mmol/kg in Contrast-enhanced 3D-Magnetic Resonance Angiography in Patients With Arterial Disease in the Abdominal to Leg Regions in the Ability of Detecting of Vessel Abnormalities
Brief Title: Magnevist (SH L 451A) Intra-individual Dose Comparison Study in Magnetic Resonance Angiography
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 91396; 308612
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2013-10-14 (Estimated); Status verified 2013-10

CONDITIONS: Magnetic Resonance Angiography; Peripheral Vascular Diseases; Peripheral Arterial Diseases
Keywords: Magnevist; Magnetic Resonance Angiography; Meglumine gadopentetate; Determination of effective dose in MRA
MeSH Terms: conditions — Peripheral Vascular Diseases; Peripheral Arterial Disease | interventions — Gadolinium DTPA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882, SH L 451A)
- Arm 2 (Experimental)
  Interventions: Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882, SH L 451A)

INTERVENTIONS:
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882, SH L 451A) — Magnevist at a dose of 0.1 mmol/kg
  Arms: Arm 1
Drug: Gadopentetate dimeglumine (Magnevist, BAY86-4882, SH L 451A) — Magnevist at a dose of 0.2 mmol/kg
  Arms: Arm 2

SUMMARY:
The objective of the study was to compare the efficacy of Magnevist (SH L 451 A) at doses of 0.1 mmol/kg and 0.2 mmol/kg in contrast-enhanced 3D-Magnetic Resonance Angiography in three regions (abdominal, femoral, and leg regions) for visualization of arteries, evaluating 179 not assessable: caused by contrast media in the evaluation of structural abnormalities. Magnevist (SH L 451 A) was administered intravenously in a crossover design in patients with arterial disease in the abdominal to leg regions. The safety of the 0.2 mmol/kg dose was also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to undergo contrast-enhanced 3D-Magnetic Resonance Angiography

Exclusion Criteria:

* Patients with an ankle brachial pressure index (ABPI) of 0.3 or less
* Patients with allergy to contrast media
* Patients with serious hepatic impairment
* Patients with serious renal impairment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2004-07; Primary Completion 2004-10 (Actual); Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
Diagnostic ability | MRI image in blinded read

SECONDARY OUTCOMES:
Visibility | MRI image in blinded read
Diagnostic confidence | MRI image in blinded read

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Japan (3):
  - Hirosaki-shi, Aomori
  - Funai-gun, Kyoto
  - Hamamatsu, Shizuoka